CLINICAL TRIAL: NCT04313452
Title: Studying the Effect of Mediterranean Diet on Insulin Resistance Compared to the Regular Diet Among Obese Children and Adolescents Aged 10-16 Years.
Brief Title: Studying the Effect of Mediterranean Diet on Insulin Resistance Among Obese Children and Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Yasmine Farrah, University of Jordan, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 8170598
Record Dates: First submitted 2020-02-24; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Obesity, Childhood; Insulin Resistance
Keywords: Mediterranean Diet
MeSH Terms: conditions — Pediatric Obesity; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: The study sample will consist of 50 participants of obese children and adolescents between 10 and 16 years of age who are diagnosed with insulin resistance clinically. Twenty five of participants (1:1, boys: girls) will follow Mediterranean diet, and 25 of participants (1:1, boys: girls) will follow regular diet. The two groups will be matched for age and gender. The Pediatric Endocrinologist will diagnose the children with insulin resistance clinically according to abdominal obesity and presence of acanthosis nigricans. The children and adolescents will be randomly assigned to one of the groups: Mediterranean diet group or the regular diet group.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- regular diet (Placebo Comparator): 50% of energy from carbohydrates, 30% fat and 20% from protein
  Interventions: Other: the effect of Mediterranean diet on insulin sensitivity among obese children and adolescents aged
- Mediterranean diet (Active Comparator): 60% of energy from carbohydrates, 25% fat and 15% from protein
  Interventions: Other: the effect of Mediterranean diet on insulin sensitivity among obese children and adolescents aged

INTERVENTIONS:
Other: the effect of Mediterranean diet on insulin sensitivity among obese children and adolescents aged — to find the effect of Mediterranean diet on insulin resistance among obese children and adolescents aged 10-16 years with insulin resistance compared to the regular diet
  Other Names: Diet intervention

SUMMARY:
Insulin resistance is a common complication of childhood obesity. It is considered to be an important link between adiposity and the risk factor of type 2 diabetes in children. The lifestyle modifications, including a healthy diet, physical activity and weight reduction in obese children and adolescents have been proven effective in type 2 diabetes prevention and management. Although increasing evidence suggests that Mediterranean diet could be associated with decreased risk of metabolic syndrome, diabetes, obesity and atherosclerosis in adults.

The importance of this study is to find the effect of Mediterranean diet on insulin resistance among obese children and adolescents aged 10-16 years. Additionally, the results of the present study will help health professionals particularly dietitians in directing children with insulin resistance towards adopting healthy diet and lifestyle.

DETAILED DESCRIPTION:
This Experimental clinical trial study will be conducted in Amman, the capital of Jordan to compare the effect of Mediterranean diet and regular diet on insulin resistance among 50 participants of obese children and adolescents (between 10 and 16 years of age) who are diagnosed with insulin resistance clinically, Twenty five of participants (1:1, boys: girls) will follow Mediterranean diet, and 25 of participants (1:1, boys: girls) will follow regular diet. The two groups will be matched for age and gender. The Pediatric Endocrinologist will diagnose the children with insulin resistance clinically according to abdominal obesity and presence of acanthosis nigricans. The children and adolescents will be randomly assigned to one of the groups: Mediterranean diet group or the regular diet group. Patients are visiting the Pediatric Diabetes and Endocrinology department in Jordan University Hospital. will be followed-up every 2 weeks in the clinic for 6 months.

The researcher will measure body weight , height, and calculate BMI for all patients every visit. Then will be represented and interpreted using the suitable growth chart (weight for age, height for age, BMI for age and gender).

Glycated hemoglobin (HbA1c), serum concentrations of total cholesterol, high-density lipoprotein (HDL) cholesterol, low-density lipoprotein (LDL) cholesterol, triglycerides, (after a 12 hour fast), aspartate aminotransferase (AST), and alanine aminotransferase (ALT), Kidney function, thyroid hormone will be recorded from the medical file of the patients.

Insulin resistance will be assessed by the homeostatic model assessment (HOMA-IR), calculated as the product of the fasting plasma insulin level (IU/l) and the fasting plasma glucose level (mmol/l) divided by 22.5. The fasting plasma insulin level (FPI) and the fasting plasma glucose level (FPG) will be measured after at least an 8-hour fasting at baseline after 3 months, and at the end of the intervention.

The intervention programs will be based on the implementation of Mediterranean diet and regular diet. Participants will be counseled and educated about the two diet programs. The two groups will be:

Group 1: regular diet ( 50% of energy from carbohydrates, 30% fat and 20% from protein) Group 2: Mediterranean diet ( 60% of energy from carbohydrates, 25% fat and 15% from protein).

ELIGIBILITY:
Inclusion Criteria:

* Age range between 10-16 years.
* Obese children and adolescents, BMI for age and sex is greater than the +2rd z-score, according to WHO growth chart.
* Children and adolescents diagnosed with insulin resistance and presence of acanthosis nigricans.
* Not on medication.

Exclusion Criteria:

* Age younger than 10 years or older than 16 years.
* Overweight children and adolescents or obese (BMI for age and sex is less than +2rd z-score, according to WHO growth chart.
* Children and adolescents didn't diagnosis of insulin resistance
* On any medication.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2020-02-27 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Mediterranean Diet and insulin Resistance | 6 month
  Mediterranean Diet change of blood level of Homa IR among Obese Children and Adolescents
Mediterranean Diet and body weight | 6 month
  Mediterranean Diet change in body weight in kilogram among Obese Children and Adolescents

SECONDARY OUTCOMES:
Mediterranean Diet and lipid profile | 6 month
  Mediterranean Diet change of blood level of lipid profile among Obese Children and Adolescents

CONTACTS AND LOCATIONS:
Overall Officials: Reema F Tayyam, PHD, Study Director — University of Jordan
Locations (1):
- University of Jordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Yes
-The study sample will consist of 50 participants of obese children and adolescents between 10 and 16 years of age who are diagnosed with insulin resistance clinically.
  Twenty five of participants (1:1, boys: girls) will follow Mediterranean diet, and 25 of participants (1:1, boys: girls) will follow regular diet. The two groups will be matched for age and gender. The Pediatric Endocrinologist will diagnose the children with insulin resistance clinically according to abdominal obesity and presence of acanthosis nigricans. The children and adolescents will be randomly assigned to one of the groups: Mediterranean diet group or the regular diet group. The study will be started after getting the Institutional Review Boards (IRB) approval.
Supporting Information: Study Protocol, CSR
Time Frame: Patients will be followed-up every 2 weeks in the clinic for 6 months
Access Criteria: Obese children and adolescents, BMI for age and sex is greater than the +2rd z-score, according to WHO growth chart, age between 10-16 years.
  Children and adolescents diagnosed with insulin resistance and presence of acanthosis nigricans and not on medication.

REFERENCES:
- [Background] Cruz ML, Weigensberg MJ, Huang TT, Ball G, Shaibi GQ, Goran MI. The metabolic syndrome in overweight Hispanic youth and the role of insulin sensitivity. J Clin Endocrinol Metab. 2004 Jan;89(1):108-13. doi: 10.1210/jc.2003-031188. PMID 14715836
- [Result] Arslanian S, Kim JY, Nasr A, Bacha F, Tfayli H, Lee S, Toledo FGS. Insulin sensitivity across the lifespan from obese adolescents to obese adults with impaired glucose tolerance: Who is worse off? Pediatr Diabetes. 2018 Mar;19(2):205-211. doi: 10.1111/pedi.12562. Epub 2017 Jul 20. PMID 28726334
- [Result] Bener A. Prevalence of obesity, overweight, and underweight in Qatari adolescents. Food Nutr Bull. 2006 Mar;27(1):39-45. doi: 10.1177/156482650602700106. PMID 16572718
- [Result] Bos MB, de Vries JH, Feskens EJ, van Dijk SJ, Hoelen DW, Siebelink E, Heijligenberg R, de Groot LC. Effect of a high monounsaturated fatty acids diet and a Mediterranean diet on serum lipids and insulin sensitivity in adults with mild abdominal obesity. Nutr Metab Cardiovasc Dis. 2010 Oct;20(8):591-8. doi: 10.1016/j.numecd.2009.05.008. Epub 2009 Aug 18. PMID 19692213
- [Result] Davis C, Bryan J, Hodgson J, Murphy K. Definition of the Mediterranean Diet; a Literature Review. Nutrients. 2015 Nov 5;7(11):9139-53. doi: 10.3390/nu7115459. PMID 26556369